CLINICAL TRIAL: NCT04803838
Title: The Gut and Oral Bacteria, Atherosclerosis and Ischemic Stroke Study
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Mona Skjelland, Clinical Professor, Oslo University Hospital
Other Study IDs: REK 2017/2202
Record Dates: First submitted 2018-09-10; First posted 2021-03-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke; Atherosclerosis; Microbiota
MeSH Terms: conditions — Ischemic Stroke; Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples Feces Saliva Carotid plaque
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patiens: Patients With symptomatic or asymptomatic carotid stenosis (> 50%, NASCET criteria)
  Interventions: Other: No intervention
- Controls: For study 1: Healthy Controls, volunters (mostly blood donors) For study 2 and 3: Spouses/someone living in the same household as the patient.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The main aim of this project is to demonstrate an association between gut and oral microbiota and their metabolites to carotid atherosclerosis and risk of ischemic stroke.

The investigators aim to show that these metabolite levels are diet-dependent (mainly egg yalk and red meat) and associated with specific types of microbiota.

The investigators to assess serum microbiota metabolite levels as a predictor of stroke and plaque progression for patients with carotid atherosclerosis.

DETAILED DESCRIPTION:
The Project will include four studies:

Study 1: (Comparative cross-sectional study) The main objective in this study is to assess if patients with carotid atherosclerosis have increased serum levels gut microbiota dependent metabolites compared to healthy controls.

This study will be done on prospectively collected information already available in our existing database. Approximately 215 patients will be included in this study where collected samples will be analyzed and levels of metabolites quantified. These metabolite levels will be compared to a control group of 70 healthy controls without carotid atherosclerosis (verified by ultrasound), cardiovascular outcome defined as stroke/TIA or vascular death, as well as traditional risk factors for ischemic stroke (diabetes, hypertension, smoking and coronary artery disease).

Study 2: (Comparative cross-sectional study) The aim of this study is to asses if microbiota and microbiota metabolite Levels are Associated With certain types of diet, in particular Rich in red meat and egg yalk.

In this study, 215 patients with ultrasound verified carotid atherosclerosis with or without symptoms of TIA/stroke will be compared to 70 controls. Dietary intake and food habits will be recorded using the SmartDiet questionnaire developed by 'Lipidklinikken Rikshospitalet'. Feces, saliva and blood will be collected analyzed for microbiota and metabolites. Antroprometrics, blood pressure and pulse will be recorded.

In patients undergoing carotid endarterectomy and immunohistochemical analysis will be done.

Study 3: (Comparative cross-sectional study) The aim of this study is to evaluate correlation between the microbiota and microbiota metabolite Levels With other inflammatory markers in blood, as well as known risk factors for stroke and inflammation on imaging modalities (ultrasound, 3-T MRI and PET/CT) .

In this study, 215 patients with ultrasound verified carotid atherosclerosis with or without symptoms of TIA/stroke will be compared to 70 controls.

Patients will undergo investigations with carotid ultrasound, carotid and cerebral MR imaging, blood tests including inflammatory biomarkers. A sub-group of patients will in addition undergo PET/CT imaging of carotid arteries.

Study 4: (Follow up study) The aim of this study is to evaluate the ability of microbiota and microbiota metabolites to predict ischemic stroke in patient With carotid stenosis.

Patients in study 2 and 3 will be followed up after 2 years with repetition of investigations. Findings with serum levels of microbiota metabolites, traditional risk factors and imaging will be correlated to clinical and radiological ischemic events and plaque progression.

ELIGIBILITY:
Inclusion Criteria:

- patients >18 years with an symptomatic og asymptomatic atherosclerotic carotid stenosis ≥ 50% (NASCET criteria)

Exclusion Criteria:

* active infection
* current antibiotic treatment
* autoimmune or autoinflammatory disease
* malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - All patients >18 years with an atherosclerotic carotid stenosis ≥ 50% admitting our department (Dep of Neurology, Rikshospitalet, OUH) as in-patient or out-patient will consecutively be considered for inclusion.
  Cooperation With Dep of vascular surgery Akershus University Hospital and Dep of vascular surgery, Aker, OUH, for patients scheduled for thrombendarterectomy.
  - Control Group: For study 1: Healthy volonteers For study 2 and 3: Spouses/partners where possible, otherwise matched for age and sex
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants With MRI-confirmed acute ischemic stroke related to increased Levels of serum microbiota-metabolites as assessed by blood tests. | 2 years
  Blood test (microbiota-metabolites e.g. TMAO) at study inclusion, carotid ultrasound (carotid plaque assessment and degree of stenosis) and cerebral MRI (evidence of stroke) at follow up

SECONDARY OUTCOMES:
Number of participants with progression of carotid stenosis related to increased Levels of serum microbiota-metabolites as assessed by blood tests. | 2 years
  Blood tests (microbiota metabolites e.g. TMAO) and carotid ultrasound (plaque assessment and degree of stenosis)
Number of participants With increased Levels of microbiota-metabolites related to Diet Rich in red meat and egg yalk as assessed by 'Smart Diet' questionnaire. | At inclusion
  Blood tests (microbiota metabolites, e.g. TMAO), dietary questionnaire ('Smart Diet' developed by the department for endocrinology Rikshospitalet)
Number of participants With increased Levels of microbiota-metabolites related to specific types of microbiota in feces and saliva as assessed by next generation sequencing and 16S RNA. | At inclusion
  Blood tests (microbiota metabolites e.g TMAO), fecal samples (Next generation sequencing, 16S RNA), saliva samples (Next generation sequencing 16S RNA)
Number of participants With increased Levels of microbiota-metabolites related to traditional risk factors for ischemic stroke assessed by questionnaire and Medical journal. | At inclusion
  Blood tests (microbiota metabolites, e.g. TMAO), questionnaire (Risk factors: hypertension, diabetes mellitus type 2, previous stroke og myocardial infarction, smoking, physical inactivity, Family history)
Number of participants With increased Levels of microbiota-metabolites related to signs of plaque instability on imaging studies assessed by carotid ultrasound, carotid and cerebral MRI and for a subgroup: carotid PET/CT. | At inclusion
  Blood tests (microbiota metabolites, e.g. TMAO), carotid ultrasound (carotid plaque assessment, degree of stenosis), carotid and cerebral MRI (evidence of inflammation and stenosis in carotids, stroke), for a subgroup: carotid PET/CT (evidence of inflammation)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided